CLINICAL TRIAL: NCT06079307
Title: Effect of Oxygenated Mouthwash and Mouth Foam on Oral Health and Quality of Life
Brief Title: Effect of Oxygenated Mouthwash and Mouth Foam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-23- KSU-1001
Record Dates: First submitted 2023-05-19; First posted 2023-10-12 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-05

CONDITIONS: Gingival Diseases; Plaque, Dental; Quality of Life
MeSH Terms: conditions — Gingival Diseases; Dental Plaque

STUDY DESIGN:
Intervention Model Description: 3 parallel arms running for 12 months and six-points data collection (examination - plaque index and gingival index)
Who Masked: Outcomes Assessor
Masking Description: due to ethical consideration participants cannot be blinded nor examiners as they will be providing oral hygiene instructions and information relative to using the mouth rinse and the mouth foam. everyone handling the data after examination will be blinded, they will be dealing with data obtained after identifying an identification code to each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Won't receive an oxygenated mouthwash nor oxygenated mouth foam yet will be provided a fluoridated toothpaste and a toothbrush (20 participants)
- Oxygenated mouthwash Group (Experimental): Provided with oxygenated mouthwash bottle 2 per individual for 3 months (40 bottles in total). -20 participants -
  Interventions: Other: Oxygenated Mouthwash
- Oxygenated mouth foam Group (Experimental): Provided with oxygenated mouth foam/ day- 20 participants- 2 oxygenated mouth foam bottle per individual for 3 months (40 bottles in total).
  Interventions: Other: Oxygenated mouth foam

INTERVENTIONS:
Other: Oxygenated Mouthwash — Will be comparing the impact of using oxygenated mouthwash with other groups.
  Arms: Oxygenated mouthwash Group
Other: Oxygenated mouth foam — will be comparing the impact of using oxygenated foam to other groups.
  Arms: Oxygenated mouth foam Group

SUMMARY:
The Aim of this independent, parallel, twelve-week clinical study is to assess the efficacy of a commercially available oxygenated mouth rinse and mouth foam on both plaque level and gingival status in addition to assessing the oral health related quality of life.

DETAILED DESCRIPTION:
Participants in all groups will be examined for gingival inflammation and plaque accumulation. The difference between three trial arms lies in the product used (control, oxygenated mouth wash, oxygenated mouth foam). A comparison against no intervention was disregarded due to ethical concerns (children only examined without informing them about their oral problems). After examination at baseline participants will be assigned to one arm of intervention. All participants will be provided an oral health education and gingival scaling to remove any underlining predisposing factor for gingival inflammation as well as fluoridated toothpaste and a toothbrush. Participants within intervention arms will also be provided the product package and informed how to use it (oxygenated mouth wash, oxygenated mouth foam).

All three arms will be followed after (1week, 2 weeks, 4 weeks, 8 weeks and 12 weeks) from baseline examination.

1. Control group Won't receive an oxygenated mouthwash nor oxygenated mouth foam (20 participants) 2. Intervention Group A: 20 participants - 2 oxygenated mouthwash bottle per individual for 3 months (40 bottles in total).

3. Intervention Group B: Oxygenated mouth foam/ day 20 participants- 2 oxygenated mouth foam bottle per individual for 3 months (40 bottles in total).

ELIGIBILITY:
Inclusion Criteria:

* Students and employees at College of applied Medical science over 19 years old
* Both Saudis and non-Saudis.
* Students and employees consenting to participate.

Exclusion Criteria:

* Intern students or students in their 1st year.
* Students and employees with medically compromised condition (including congenital heart disease, hematological condition, immune deficiency condition and end stage renal disease or those with organ transplant within the previous 5 year.
* Students and employees not consenting to participate.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Gingival index | baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Gingival index | +1 week from baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Gingival index | +2 weeks from baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Gingival index | +4 weeks from baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Gingival index | +8 weeks from baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Gingival index | +12 weeks from baseline
  Gingival index has been used to clinically characterize the degree of gingival inflammation. were the scale range 0-3. zero indicating the best results and 3 as sever gingivitis.
Plaque index | baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation.
Plaque index | +1 week from baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation
Plaque index | +2 weeks from baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation
Plaque index | +4 weeks from baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation
Plaque index | +8 weeks from baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation
Plaque index | +12 weeks from baseline
  Oral hygiene may be assessed via a plaque index also plaque is a predisposing factor for gingival inflammation

SECONDARY OUTCOMES:
Gum Health Experience Questionnaire (GHEQ) | Baseline
  The questions are designed to assess the impact that gum-related symptoms may have on your everyday life. (Assessed through Likert scale were the 5 is the highest score and 1 is the lowest score)
Gum Health Experience Questionnaire (GHEQ) | +12 weeks from baseline
  The questions are designed to assess the impact that gum-related symptoms may have on your everyday life. (Assessed through Likert scale were the 5 is the highest score and 1 is the lowest score)

CONTACTS AND LOCATIONS:
Overall Officials: Haya M Alayadi, PhD, Principal Investigator — King Saud University
Locations (1):
- Haya Mahmmod Alayadi, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The principle investigator will be responsible for all data entry and management. Personal identification will be collected to regain contact with participants for the follow-up assessments and link baseline with follow-up data. This will be handled through pseudo anonymization, whereby the principle investigator will keep a separate file containing personal identifiable information for all participants and assign an identification code to each as they enter the study. Other than the examiner in the clinic everybody else will be working with coded data when analyzing the information.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: upon the completion of the trial
Access Criteria: study protocol as well as statistical analysis plane will be shared through a published paper as well as reporting back to trials.gov and clinical study report will be shared through trials.gov

REFERENCES:
- [Background] Allen F, Locker D. A modified short version of the oral health impact profile for assessing health-related quality of life in edentulous adults. Int J Prosthodont. 2002 Sep-Oct;15(5):446-50. PMID 12375458
- [Background] Ciancio SG. Current status of indices of gingivitis. J Clin Periodontol. 1986 May;13(5):375-8, 381-2. doi: 10.1111/j.1600-051x.1986.tb01476.x. PMID 3522646
- [Background] Fischman SL. Current status of indices of plaque. J Clin Periodontol. 1986 May;13(5):371-4, 379-80. doi: 10.1111/j.1600-051x.1986.tb01475.x. PMID 3013947
- [Background] Broomhead T, Gibson BJ, Parkinson C, Robinson PG, Vettore MV, Baker SR. Development and psychometric validation of the gum health experience questionnaire. J Clin Periodontol. 2024 Jan;51(1):33-42. doi: 10.1111/jcpe.13878. Epub 2023 Sep 21. PMID 37735867
- [Background] Broomhead T, Gibson B, Parkinson CR, Vettore MV, Baker SR. Gum health and quality of life-subjective experiences from across the gum health-disease continuum in adults. BMC Oral Health. 2022 Nov 18;22(1):512. doi: 10.1186/s12903-022-02507-5. PMID 36401324